CLINICAL TRIAL: NCT06958302
Title: The Relation Between Diabetic Neuropathy and Muscle Mass in Type 2 Diabetes Mellitus Patients
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD16/2025
Record Dates: First submitted 2025-04-06; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Neuropathy; Sarcopenia
Keywords: diabetic neuropathy; muscle mass; sarcopenia; nerve conduction studies
MeSH Terms: conditions — Diabetic Neuropathies; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- type 2 diabetic patients: type 2 diabetes mellitus patients aged above 45 years old and tested for diabetic neuropathy

SUMMARY:
The goal of this observational study is to evaluate the relation between diabetic neuropathy in type 2 diabetes mellitus patients and muscle mass

DETAILED DESCRIPTION:
The goal of this observational study is to evaluate the relation between diabetic neuropathy in type 2 diabetes mellitus patients, aged above 45 years old, and muscle mass; where it uses ultrasound to measure anterior thigh muscle thickness and adjusts it to body mass index to calculate muscle mass and the participants perform clinical tests i.e hand grip strength test and chair stand test in order to assess muscle power. Depending on both muscle mass and muscle power/function, Sarcopenia could be assessed in this group of patients, and its relation to diabetic neuropathy, tested by nerve conduction studies, would be researched.

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of patients diagnosed with Type 2 diabetes mellitus aged ≥45 years old

Exclusion Criteria:

* Type 1 DM, gestational diabetes mellitus
* Severe cardiopulmonary disease, significant/previous neurological disorder (e.g., ischemic stroke, Parkinson disease) causing difficulty during daily activities (e.g., walking), visual deficit, and psychiatric problem
* Other neuropathy-associated factors such as: alcohol, nutrition, poisoning and drug addiction
* Patients with renal diseases, malignancy and autoimmune diseases
* Patients on long term use of Steroids

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group consisted of patients diagnosed with Type 2 diabetes mellitus aged ≥45 years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Relation between diabetic neuropathy and muscle mass | Day 1 Neurological examination and clinical physical performance tests for sarcopenia, 2 weeks later: nerve conduction studies for both lower limbs, the 3rd week: ultrasound assessment for thigh muscle thickness
  Relation between Diabetic neuropathy severity (mild/moderate/severe) using nerve conduction studies classification criteria (Baba's classification) and skeletal muscle mass as indicated by a ratio (anterior thigh muscle thickness measured by ultrasound/ BMI) (millimeteres for muscle thickness ) and (kg/m^2 for the BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Rana A Al Hilaly, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kara M, Kaymak B, Frontera W, Ata AM, Ricci V, Ekiz T, Chang KV, Han DS, Michail X, Quittan M, Lim JY, Bean JF, Franchignoni F, Ozcakar L. Diagnosing sarcopenia: Functional perspectives and a new algorithm from the ISarcoPRM. J Rehabil Med. 2021 Jun 21;53(6):jrm00209. doi: 10.2340/16501977-2851. PMID 34121127
- [Background] Perkisas S, Baudry S, Bauer J, Beckwee D, De Cock AM, Hobbelen H, Jager-Wittenaar H, Kasiukiewicz A, Landi F, Marco E, Merello A, Piotrowicz K, Sanchez E, Sanchez-Rodriguez D, Scafoglieri A, Cruz-Jentoft A, Vandewoude M. Application of ultrasound for muscle assessment in sarcopenia: towards standardized measurements. Eur Geriatr Med. 2018 Dec;9(6):739-757. doi: 10.1007/s41999-018-0104-9. Epub 2018 Sep 17. PMID 34674473
- [Background] Pinheiro PA, Carneiro JA, Coqueiro RS, Pereira R, Fernandes MH. "Chair Stand Test" as Simple Tool for Sarcopenia Screening in Elderly Women. J Nutr Health Aging. 2016 Jan;20(1):56-9. doi: 10.1007/s12603-016-0676-3. PMID 26728934
- [Background] Bohannon RW. Test-Retest Reliability of Measurements of Hand-Grip Strength Obtained by Dynamometry from Older Adults: A Systematic Review of Research in the PubMed Database. J Frailty Aging. 2017;6(2):83-87. doi: 10.14283/jfa.2017.8. PMID 28555708
- [Background] Kara M, Kaymak B, Ata AM, Ozkal O, Kara O, Baki A, Sengul Aycicek G, Topuz S, Karahan S, Soylu AR, Cakir B, Halil M, Ozcakar L. STAR-Sonographic Thigh Adjustment Ratio: A Golden Formula for the Diagnosis of Sarcopenia. Am J Phys Med Rehabil. 2020 Oct;99(10):902-908. doi: 10.1097/PHM.0000000000001439. PMID 32941253
- [Background] Tsukasaki K, Matsui Y, Arai H, Harada A, Tomida M, Takemura M, Otsuka R, Ando F, Shimokata H. Association of Muscle Strength and Gait Speed with Cross-Sectional Muscle Area Determined by Mid-Thigh Computed Tomography - A Comparison with Skeletal Muscle Mass Measured by Dual-Energy X-Ray Absorptiometry. J Frailty Aging. 2020;9(2):82-89. doi: 10.14283/jfa.2020.16. PMID 32259181
- [Background] Abe T, Loenneke JP, Thiebaud RS, Ogawa M, Mitsukawa N. Age-related site-specific muscle loss in the thigh and zigzag walking performance in older men and women. Acta Physiol Hung. 2014 Dec;101(4):488-95. doi: 10.1556/APhysiol.101.2014.006. PMID 25201711
- [Background] Ata AM, Kara M, Kaymak B, Gurcay E, Cakir B, Unlu H, Akinci A, Ozcakar L. Regional and total muscle mass, muscle strength and physical performance: The potential use of ultrasound imaging for sarcopenia. Arch Gerontol Geriatr. 2019 Jul-Aug;83:55-60. doi: 10.1016/j.archger.2019.03.014. Epub 2019 Mar 19. PMID 30953961
- [Background] Chen F, Xu S, Wang Y, Chen F, Cao L, Liu T, Huang T, Wei Q, Ma G, Zhao Y, Wang D. Risk Factors for Sarcopenia in the Elderly with Type 2 Diabetes Mellitus and the Effect of Metformin. J Diabetes Res. 2020 Oct 7;2020:3950404. doi: 10.1155/2020/3950404. eCollection 2020. PMID 33083494